CLINICAL TRIAL: NCT05684367
Title: Center-Based and Home-Based Walking Exercise Intervention to Reduce Fatigue in Older Breast Cancer Survivors
Brief Title: Exercise to ReGain Stamina and Energy (The EXERGISE Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202202679; OCR42286 (Other: UF OnCore); IRB202102537 (Other: UF)
Record Dates: First submitted 2022-08-23; First posted 2023-01-13 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Fatigue; Breast Cancer; Cancer, Therapy-Related
MeSH Terms: conditions — Fatigue; Breast Neoplasms; Neoplasms, Second Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Center-Based Walking Exercise (Experimental): Subjects will be randomly assigned to receive a center-based walking exercise intervention 3 days per week for the duration of the study.
  Interventions: Behavioral: Center-Based Walking Exercise
- Home-Based Walking Exercise (Experimental): Subjects will be randomly assigned to walk for exercise in their community five days/week.
  Interventions: Behavioral: Home-Based Walking Exercise

INTERVENTIONS:
Behavioral: Center-Based Walking Exercise — Each exercise session will begin with a short warm-up followed by 30 min of walking. Participants will initially be instructed to walk at a moderate intensity, equivalent to a 5-6 on Borg category-ratio (CR) scale. Participants will be encouraged to, if possible, incorporate brief periods of vigorous walking (7-8 on CR10 scale) with a goal of achieving at least 10 min of vigorous walking per session.
  Arms: Center-Based Walking Exercise
Behavioral: Home-Based Walking Exercise — Participants will be asked to walk for exercise in their community five days/week. Participants will be instructed to begin with 10-15 minutes of walking exercise/session in the first month of the intervention and to increase exercise duration by five minutes/session each week, facilitating reasonable but steady progress toward the goal of 30 minutes per session.
  Arms: Home-Based Walking Exercise

SUMMARY:
About 20%-70% of breast cancer survivors experience fatigue after cancer therapy. Because epidemiologic evidence shows that old age is a risk factor for fatigue in adults with cancer history, older breast cancer survivors suffer from even more fatigue than younger survivors. The purpose of this study is to test types of walking exercise interventions and their ability to reduce fatigue in older breast cancer survivors.

DETAILED DESCRIPTION:
Women with breast cancer often experience severe fatigue (asthenia) after cancer therapy, seen in approximately 40% of breast cancer survivors. Because older age is a risk factor for fatigue, older breast cancer survivors are at an increased risk versus those in younger age groups. Prior evidence suggests that aerobic exercise reduces inflammation and bioenergenesis disturbance, which are key factors that drive the pathogenesis of fatigue. Although interventional studies suggest that aerobic exercise can improve fatigue in younger breast cancer survivors, anti-fatigue effects of aerobic exercise tended to decrease with increasing age. The investigators postulate that novel interventions combined with aerobic exercise can enhance its effectiveness and alleviate severe fatigue further in older breast cancer survivors.

In this pilot randomized clinical trial, the investigators will enroll 24 female cancer survivors aged ≥ 60 years who were diagnosed with invasive breast cancer but have completed adjuvant therapy for at least 3 months but no more than 1 year. Participants will be randomly assigned to either a center-based walking exercise intervention or a home-based walking exercise intervention for an 8 week period. By completing this pilot study, the investigators will be able to collect preliminary data; refine the recruitment, measurement, randomization, and retention strategy; and adjust the statistical strategy and timeline for the potential full-scale randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate in the study
* Age ≥ 60 years old
* Had stage I-III invasive breast cancer
* The cancer is diagnosed in 2021 or 2022
* Completed adjuvant therapy for at least 3 months but no more than 1 year
* Willingness to participate in all study procedures
* Had at least moderate-level fatigue (defined as raw score ≥ 8 on the PROMIS Measure)

Exclusion Criteria:

* Failure to provide informed consent
* Current involvement in rehabilitation program
* Absolute contraindications to exercise training
* Significant cognitive impairment
* Progressive, degenerative neurologic disease
* Hip fracture, hip or knee replacement, or spinal surgery within past 4 months
* Other significant comorbidities that may impair ability to participate in the exercise intervention
* Pregnant
* Regular consumption of nicotinamide riboside supplement
* Simultaneous participation in other interventional studies
* Had no or very mild fatigue (defined as raw score ≤7 in PROMIS)
* Diagnosis of any of the following medical conditions in past three years (coronary heart disease, angina, heart attack, heart failure, stroke, high blood pressure, chronic obstructive pulmonary disease, chronic bronchitis, arthritis, diabetes mellitus, and chronic kidney disease), as measured by Behavioral Risk Factor Surveillance System
* Receipt of any oral or intravenous antibiotic 4 weeks prior to screening
* Receipt of any probiotics within 4 weeks of screening
* History of active treatment for HIV, hepatitis B, or hepatitis C infection
* Positive stool cultures for enteric pathogens, including Clostridium difficile
* Excessive alcohol use (i.e., > 14 drinks/week) or alcohol abuse (i.e., > 5 drinks/day for males or > 4 drinks/day for females)
* Other substance abuse within the past 3 years
* Smoking history in past 3 years

Ages: 60 Years to 105 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Because the study population will be older (60+ years) breast cancer survivors, only women will be enrolled in this pilot study. Although men can also have breast cancer, the risk is extremely low (ratio of male vs. female incident breast cancer = 1:100), thus the study does not consider men in this pilot study.
Enrollment: 24 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Self-Reported Fatigue | Baseline up to Week 8
  Patient Reported Outcomes Measurement Information System (PROMIS) is a set of person-centered measures that evaluate and monitor physical, psychological, and social health based on experts' review of items reflecting general health, functional status, and quality of life. All items are measured based on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) and PROMIS reverse scores item 7. Scores of all items are summed, with higher scores indicating greater fatigue. Raw total scores will range from 7 to 35.

SECONDARY OUTCOMES:
Mental Distress (Depression and Anxiety) | Baseline up to Week 8
  Mental distress (depression and anxiety) in past 7 days will be measured by PROMIS. Participants will answer 8 and 7 questions to reflect severity of depression and anxiety, respectively; for each question, a 5-point scale and normalized T-scores will be employed as measure of fatigue.
Self-Reported Pain | Baseline up to Week 8
  Self-reported pain in past 7 days will be measured by 6 questions in PROMIS Pain Interference Short Form; the questions measure severity of pain and use a 5-point scale (1=not at all; 2=a little bit; 3=somewhat; 4=quite a bit; 5=very much) whose sum can be transformed to a normalized T-score.
Self-Reported Sleep Disturbance | Baseline up to Week 8
  Self-reported sleep short form (8a) that assesses the pure domain of sleep disturbance in individuals aged 18 and older. Each item on the measure is rated on a 5-point scale (1=very good; 2=good; 3=fair; 4=poor; and 5=very poor) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance whose sum can be transformed to a normalized T-score.
Gait Speed | Baseline up to Week 8
  Gait speed will be assessed in by the 6 Minute Walk test, which measures the amount of distance the participant can complete on a standard walking course in six minutes without running or overexerting themselves. Gait speed will be measured by approach used in the National Health and Nutrition Examination Survey; participants will be asked to finish a 20-foot walking test and gait speed will be calculated as (20×0.3048 meter)/(time (seconds) to finish test).
Physical Function | Baseline up to Week 8
  Physical function will be assessed by the the Short Physical Performance Battery (SPPB). This battery assess functional performance on different tasks including timed short distance walk, repeated chair stands, and a balance test. Additionally, isometric grip strength, a commonly used measure of upper body skeletal function, will be assess with a hand held dynamometer.
Treatment-Induced Peripheral Neuropathy (TIPN) | Baseline up to Week 8
  The 10-item Treatment-induced Neuropathy Assessment Scale (TNAS) will be used to evaluate the severity and impact of peripheral neuropathy on daily functioning at baseline and following or during after chemotherapy treatment. All items are measured based on a 10-point scale. Scores of all items are summed, with higher scores indicating greater neuropathy. Two subscale scores will be calculated to evaluate symptoms related to sensory or interference dimensions. Sensory subscale score will be the mean of 6 sensory items: numbness, tingling, pain, hot or burning, feelings of coldness and disturbed sleep. The interference subscale score - the mean of 3 interference items: trouble walking, trouble with balance and difficulty using hands.
Habitual Physical Activity | Baseline up to Week 8
  Self-administered questionnaire to assess habitual physical activity through three components: work activity, sport activity, and leisure activity. The Modified Baecke Questionnaire measures habitual activity in older adults, which includes questions on household activities, sports and leisure time activities. Free-living physical activity at baseline and follow-up will be measured using an Apple Watch. Adherence to walking exercise intervention will be measured based on four criteria: total walking minutes, total walking minutes within assigned target heart rate zone, percentage of prescribed walking minutes completed per week, and percentage of prescribed walking minutes within the target heart rate zone per week.
Functional Assessment of Cancer Therapy - Breast (FACT-B) | Baseline up to Week 8
  The FACT-B is a 37-item instrument designed to measure five domains of HRQOL in breast cancer survivors: Physical, social, emotional, functional well-being as well as a breast-cancer subscale (BCS). Each item on the measure is rated on a 5 point Likert-type scale (Not at all; A little bit; Somewhat; Quite a bit; and very much).
Perceived Stress | Baseline up to Week 8
  The Perceived Stress Scale (PSS-10) covers feelings and current life situation, both of which are measured on a 5-point Likert scale (0 = never, 1 = almost never, 2 = sometimes, 3 = fairly often, 4 = very often); higher scores indicate higher perceived stress.
Dispositional Gratitude | Baseline up to Week 8
  The Gratitude Questionnaire-6 (GQ-6) is designed to measure four facets of dispositional gratitude: (a) intensity, (b) frequency, (c) span and (d) density. Each item is rated on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree). Scores range from 6 to 42, with higher scores implying a greater level of dispositional gratitude and lower scores indicating a decreased disposition in gratitude.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Anton, Principal Investigator — University of Florida
Locations (1):
- Institute on Aging; University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin CB, Herrick KA, Sarafrazi N, Ogden CL. Attempts to Lose Weight Among Adults in the United States, 2013-2016. NCHS Data Brief. 2018 Jul;(313):1-8. PMID 30044214
- [Background] Demb J, Abraham L, Miglioretti DL, Sprague BL, O'Meara ES, Advani S, Henderson LM, Onega T, Buist DSM, Schousboe JT, Walter LC, Kerlikowske K, Braithwaite D; Breast Cancer Surveillance Consortium. Screening Mammography Outcomes: Risk of Breast Cancer and Mortality by Comorbidity Score and Age. J Natl Cancer Inst. 2020 Jun 1;112(6):599-606. doi: 10.1093/jnci/djz172. PMID 31593591
- [Background] Hamer J, McDonald R, Zhang L, Verma S, Leahey A, Ecclestone C, Bedard G, Pulenzas N, Bhatia A, Chow R, DeAngelis C, Ellis J, Rakovitch E, Lee J, Chow E. Quality of life (QOL) and symptom burden (SB) in patients with breast cancer. Support Care Cancer. 2017 Feb;25(2):409-419. doi: 10.1007/s00520-016-3417-6. Epub 2016 Sep 30. PMID 27696078
- [Background] Phillips RO. A review of definitions of fatigue - And a step towards a whole definition. Transport Res F-Traf. 2015;29:48-56.
- [Background] Campos MPO, Hassan BJ, Riechelmann R, Del Giglio A. Cancer-related fatigue: a practical review. Ann Oncol. 2011 Jun;22(6):1273-1279. doi: 10.1093/annonc/mdq458. Epub 2011 Feb 16. PMID 21325448
- [Background] Fu OS, Crew KD, Jacobson JS, Greenlee H, Yu G, Campbell J, Ortiz Y, Hershman DL. Ethnicity and persistent symptom burden in breast cancer survivors. J Cancer Surviv. 2009 Dec;3(4):241-50. doi: 10.1007/s11764-009-0100-7. Epub 2009 Oct 27. PMID 19859813
- [Background] Abrahams HJG, Gielissen MFM, Schmits IC, Verhagen CAHHVM, Rovers MM, Knoop H. Risk factors, prevalence, and course of severe fatigue after breast cancer treatment: a meta-analysis involving 12 327 breast cancer survivors. Ann Oncol. 2016 Jun;27(6):965-974. doi: 10.1093/annonc/mdw099. Epub 2016 Mar 2. PMID 26940687
- [Background] Bower JE, Ganz PA, Desmond KA, Rowland JH, Meyerowitz BE, Belin TR. Fatigue in breast cancer survivors: occurrence, correlates, and impact on quality of life. J Clin Oncol. 2000 Feb;18(4):743-53. doi: 10.1200/JCO.2000.18.4.743. PMID 10673515
- [Background] Vasbinder A, Reding KW, Wang D, Han CJ, Zaslavsky O, Langford D, Cespedes Feliciano EM, Barrington WE, Paskett ED. Postdiagnosis Physical Activity: Association With Long-Term Fatigue and Sleep Disturbance in Older Adult Breast Cancer Survivors. Clin J Oncol Nurs. 2020 Aug 1;24(4):381-391. doi: 10.1188/20.CJON.381-391. PMID 32678375
- [Background] Butt Z, Rao AV, Lai JS, Abernethy AP, Rosenbloom SK, Cella D. Age-associated differences in fatigue among patients with cancer. J Pain Symptom Manage. 2010 Aug;40(2):217-23. doi: 10.1016/j.jpainsymman.2009.12.016. Epub 2010 Jun 11. PMID 20541901
- [Background] Egerton T. Self-reported aging-related fatigue: a concept description and its relevance to physical therapist practice. Phys Ther. 2013 Oct;93(10):1403-13. doi: 10.2522/ptj.20130011. Epub 2013 May 23. PMID 23704037
- [Background] Zengarini E, Ruggiero C, Perez-Zepeda MU, Hoogendijk EO, Vellas B, Mecocci P, Cesari M. Fatigue: Relevance and implications in the aging population. Exp Gerontol. 2015 Oct;70:78-83. doi: 10.1016/j.exger.2015.07.011. Epub 2015 Jul 17. PMID 26190478
- [Background] Bardwell WA, Ancoli-Israel S. Breast Cancer and Fatigue. Sleep Med Clin. 2008 Mar;3(1):61-71. doi: 10.1016/j.jsmc.2007.10.011. PMID 18769530
- [Background] Abrahams HJG, Gielissen MFM, Verhagen CAHHVM, Knoop H. The relationship of fatigue in breast cancer survivors with quality of life and factors to address in psychological interventions: A systematic review. Clin Psychol Rev. 2018 Jul;63:1-11. doi: 10.1016/j.cpr.2018.05.004. Epub 2018 May 17. PMID 29852324
- [Background] Garabeli Cavalli Kluthcovsky AC, Urbanetz AA, de Carvalho DS, Pereira Maluf EM, Schlickmann Sylvestre GC, Bonatto Hatschbach SB. Fatigue after treatment in breast cancer survivors: prevalence, determinants and impact on health-related quality of life. Support Care Cancer. 2012 Aug;20(8):1901-9. doi: 10.1007/s00520-011-1293-7. Epub 2011 Oct 13. PMID 21994001
- [Background] Galiano-Castillo N, Ariza-Garcia A, Cantarero-Villanueva I, Fernandez-Lao C, Diaz-Rodriguez L, Arroyo-Morales M. Depressed mood in breast cancer survivors: associations with physical activity, cancer-related fatigue, quality of life, and fitness level. Eur J Oncol Nurs. 2014 Apr;18(2):206-10. doi: 10.1016/j.ejon.2013.10.008. Epub 2013 Nov 5. PMID 24201014
- [Background] Avlund K. Fatigue in older adults: an early indicator of the aging process? Aging Clin Exp Res. 2010 Apr;22(2):100-15. doi: 10.1007/BF03324782. PMID 20440097
- [Background] Campisi J, d'Adda di Fagagna F. Cellular senescence: when bad things happen to good cells. Nat Rev Mol Cell Biol. 2007 Sep;8(9):729-40. doi: 10.1038/nrm2233. PMID 17667954
- [Background] Franceschi C, Garagnani P, Parini P, Giuliani C, Santoro A. Inflammaging: a new immune-metabolic viewpoint for age-related diseases. Nat Rev Endocrinol. 2018 Oct;14(10):576-590. doi: 10.1038/s41574-018-0059-4. PMID 30046148
- [Background] Imai S. The NAD World: a new systemic regulatory network for metabolism and aging--Sirt1, systemic NAD biosynthesis, and their importance. Cell Biochem Biophys. 2009;53(2):65-74. doi: 10.1007/s12013-008-9041-4. PMID 19130305
- [Background] Mills PJ, Ancoli-Israel S, Parker B, Natarajan L, Hong S, Jain S, Sadler GR, von Kanel R. Predictors of inflammation in response to anthracycline-based chemotherapy for breast cancer. Brain Behav Immun. 2008 Jan;22(1):98-104. doi: 10.1016/j.bbi.2007.07.001. Epub 2007 Aug 15. PMID 17706918
- [Background] Gallicchio L, Gadalla SM, Murphy JD, Simonds NI. The Effect of Cancer Treatments on Telomere Length: A Systematic Review of the Literature. J Natl Cancer Inst. 2018 Oct 1;110(10):1048-1058. doi: 10.1093/jnci/djy189. PMID 30272225
- [Background] Guigni BA, Callahan DM, Tourville TW, Miller MS, Fiske B, Voigt T, Korwin-Mihavics B, Anathy V, Dittus K, Toth MJ. Skeletal muscle atrophy and dysfunction in breast cancer patients: role for chemotherapy-derived oxidant stress. Am J Physiol Cell Physiol. 2018 Nov 1;315(5):C744-C756. doi: 10.1152/ajpcell.00002.2018. Epub 2018 Sep 12. PMID 30207784
- [Background] Bower JE, Lamkin DM. Inflammation and cancer-related fatigue: mechanisms, contributing factors, and treatment implications. Brain Behav Immun. 2013 Mar;30 Suppl(0):S48-57. doi: 10.1016/j.bbi.2012.06.011. Epub 2012 Jul 6. PMID 22776268
- [Background] Bower JE. Fatigue, brain, behavior, and immunity: summary of the 2012 Named Series on fatigue. Brain Behav Immun. 2012 Nov;26(8):1220-3. doi: 10.1016/j.bbi.2012.08.009. Epub 2012 Aug 31. PMID 22964543
- [Background] Rock CL, Doyle C, Demark-Wahnefried W, Meyerhardt J, Courneya KS, Schwartz AL, Bandera EV, Hamilton KK, Grant B, McCullough M, Byers T, Gansler T. Nutrition and physical activity guidelines for cancer survivors. CA Cancer J Clin. 2012 Jul-Aug;62(4):243-74. doi: 10.3322/caac.21142. Epub 2012 Apr 26. PMID 22539238
- [Background] Carteron L, Patet C, Solari D, Messerer M, Daniel RT, Eckert P, Meuli R, Oddo M. Non-Ischemic Cerebral Energy Dysfunction at the Early Brain Injury Phase following Aneurysmal Subarachnoid Hemorrhage. Front Neurol. 2017 Jul 10;8:325. doi: 10.3389/fneur.2017.00325. eCollection 2017. PMID 28740479
- [Background] Runowicz CD, Leach CR, Henry NL, Henry KS, Mackey HT, Cowens-Alvarado RL, Cannady RS, Pratt-Chapman ML, Edge SB, Jacobs LA, Hurria A, Marks LB, LaMonte SJ, Warner E, Lyman GH, Ganz PA. American Cancer Society/American Society of Clinical Oncology Breast Cancer Survivorship Care Guideline. CA Cancer J Clin. 2016 Jan-Feb;66(1):43-73. doi: 10.3322/caac.21319. Epub 2015 Dec 7. PMID 26641959
- [Background] Zhang D, Zhao Y, Kaushiva A, Zhu Z, Wang JH, Braithwaite D. Self-rated health in relation to fruit and vegetable consumption and physical activity among older cancer survivors. Support Care Cancer. 2021 May;29(5):2713-2722. doi: 10.1007/s00520-020-05782-6. Epub 2020 Sep 26. PMID 32979089
- [Background] Vieira RP, Claudino RC, Duarte AC, Santos AB, Perini A, Faria Neto HC, Mauad T, Martins MA, Dolhnikoff M, Carvalho CR. Aerobic exercise decreases chronic allergic lung inflammation and airway remodeling in mice. Am J Respir Crit Care Med. 2007 Nov 1;176(9):871-7. doi: 10.1164/rccm.200610-1567OC. Epub 2007 Aug 9. PMID 17690332
- [Background] Kuphal KE, Fibuch EE, Taylor BK. Extended swimming exercise reduces inflammatory and peripheral neuropathic pain in rodents. J Pain. 2007 Dec;8(12):989-97. doi: 10.1016/j.jpain.2007.08.001. Epub 2007 Sep 24. PMID 17890162
- [Background] Denham J, O'Brien BJ, Charchar FJ. Telomere Length Maintenance and Cardio-Metabolic Disease Prevention Through Exercise Training. Sports Med. 2016 Sep;46(9):1213-37. doi: 10.1007/s40279-016-0482-4. PMID 26914269
- [Background] Kinney LaPier TL, Rodnick KJ. Effects of aerobic exercise on energy metabolism in the hypertensive rat heart. Phys Ther. 2001 Apr;81(4):1006-17. PMID 11276183
- [Background] Arikawa AY, Thomas W, Schmitz KH, Kurzer MS. Sixteen weeks of exercise reduces C-reactive protein levels in young women. Med Sci Sports Exerc. 2011 Jun;43(6):1002-9. doi: 10.1249/MSS.0b013e3182059eda. PMID 21085036
- [Background] Zheng G, Qiu P, Xia R, Lin H, Ye B, Tao J, Chen L. Effect of Aerobic Exercise on Inflammatory Markers in Healthy Middle-Aged and Older Adults: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Front Aging Neurosci. 2019 Apr 26;11:98. doi: 10.3389/fnagi.2019.00098. eCollection 2019. PMID 31080412
- [Background] Puterman E, Weiss J, Lin J, Schilf S, Slusher AL, Johansen KL, Epel ES. Aerobic exercise lengthens telomeres and reduces stress in family caregivers: A randomized controlled trial - Curt Richter Award Paper 2018. Psychoneuroendocrinology. 2018 Dec;98:245-252. doi: 10.1016/j.psyneuen.2018.08.002. Epub 2018 Aug 2. PMID 30266522
- [Background] Hargreaves M, Spriet LL. Skeletal muscle energy metabolism during exercise. Nat Metab. 2020 Sep;2(9):817-828. doi: 10.1038/s42255-020-0251-4. Epub 2020 Aug 3. PMID 32747792
- [Background] Lahart IM, Metsios GS, Nevill AM, Carmichael AR. Physical activity for women with breast cancer after adjuvant therapy. Cochrane Database Syst Rev. 2018 Jan 29;1(1):CD011292. doi: 10.1002/14651858.CD011292.pub2. PMID 29376559
- [Background] Frasca D, Blomberg BB, Paganelli R. Aging, Obesity, and Inflammatory Age-Related Diseases. Front Immunol. 2017 Dec 7;8:1745. doi: 10.3389/fimmu.2017.01745. eCollection 2017. PMID 29270179
- [Background] Roberts SB, Rosenberg I. Nutrition and aging: changes in the regulation of energy metabolism with aging. Physiol Rev. 2006 Apr;86(2):651-67. doi: 10.1152/physrev.00019.2005. PMID 16601270
- [Background] Trammell SA, Yu L, Redpath P, Migaud ME, Brenner C. Nicotinamide Riboside Is a Major NAD+ Precursor Vitamin in Cow Milk. J Nutr. 2016 May;146(5):957-63. doi: 10.3945/jn.116.230078. Epub 2016 Apr 6. PMID 27052539
- [Background] Joshi U, Evans JE, Pearson A, Saltiel N, Cseresznye A, Darcey T, Ojo J, Keegan AP, Oberlin S, Mouzon B, Paris D, Klimas N, Sullivan K, Mullan M, Crawford F, Abdullah L. Targeting sirtuin activity with nicotinamide riboside reduces neuroinflammation in a GWI mouse model. Neurotoxicology. 2020 Jul;79:84-94. doi: 10.1016/j.neuro.2020.04.006. Epub 2020 Apr 25. PMID 32343995
- [Background] Elhassan YS, Kluckova K, Fletcher RS, Schmidt MS, Garten A, Doig CL, Cartwright DM, Oakey L, Burley CV, Jenkinson N, Wilson M, Lucas SJE, Akerman I, Seabright A, Lai YC, Tennant DA, Nightingale P, Wallis GA, Manolopoulos KN, Brenner C, Philp A, Lavery GG. Nicotinamide Riboside Augments the Aged Human Skeletal Muscle NAD+ Metabolome and Induces Transcriptomic and Anti-inflammatory Signatures. Cell Rep. 2019 Aug 13;28(7):1717-1728.e6. doi: 10.1016/j.celrep.2019.07.043. PMID 31412242
- [Background] Sun C, Wang K, Stock AJ, Gong Y, Demarest TG, Yang B, Giri N, Harrington L, Alter BP, Savage SA, Bohr VA, Liu Y. Re-equilibration of imbalanced NAD metabolism ameliorates the impact of telomere dysfunction. EMBO J. 2020 Nov 2;39(21):e103420. doi: 10.15252/embj.2019103420. Epub 2020 Sep 16. PMID 32935380
- [Background] Demaria M, O'Leary MN, Chang J, Shao L, Liu S, Alimirah F, Koenig K, Le C, Mitin N, Deal AM, Alston S, Academia EC, Kilmarx S, Valdovinos A, Wang B, de Bruin A, Kennedy BK, Melov S, Zhou D, Sharpless NE, Muss H, Campisi J. Cellular Senescence Promotes Adverse Effects of Chemotherapy and Cancer Relapse. Cancer Discov. 2017 Feb;7(2):165-176. doi: 10.1158/2159-8290.CD-16-0241. Epub 2016 Dec 15. PMID 27979832
- [Background] Dollerup OL, Christensen B, Svart M, Schmidt MS, Sulek K, Ringgaard S, Stodkilde-Jorgensen H, Moller N, Brenner C, Treebak JT, Jessen N. A randomized placebo-controlled clinical trial of nicotinamide riboside in obese men: safety, insulin-sensitivity, and lipid-mobilizing effects. Am J Clin Nutr. 2018 Aug 1;108(2):343-353. doi: 10.1093/ajcn/nqy132. PMID 29992272
- [Background] Koltai E, Szabo Z, Atalay M, Boldogh I, Naito H, Goto S, Nyakas C, Radak Z. Exercise alters SIRT1, SIRT6, NAD and NAMPT levels in skeletal muscle of aged rats. Mech Ageing Dev. 2010 Jan;131(1):21-8. doi: 10.1016/j.mad.2009.11.002. Epub 2009 Nov 12. PMID 19913571
- [Background] Pereira PTVT, Reis AD, Diniz RR, Lima FA, Leite RD, da Silva MCP, Guerra RNM, de Moraes Vieira EB, Garcia JBS. Dietary supplements and fatigue in patients with breast cancer: a systematic review. Breast Cancer Res Treat. 2018 Oct;171(3):515-526. doi: 10.1007/s10549-018-4857-0. Epub 2018 Jun 18. PMID 29915949
- [Background] Lee HJ, Yang SJ. Supplementation with Nicotinamide Riboside Reduces Brain Inflammation and Improves Cognitive Function in Diabetic Mice. Int J Mol Sci. 2019 Aug 27;20(17):4196. doi: 10.3390/ijms20174196. PMID 31461911
- [Background] Wharton S, Astrup A, Endahl L, Lean MEJ, Satylganova A, Skovgaard D, Wadden TA, Wilding JPH. Estimating and reporting treatment effects in clinical trials for weight management: using estimands to interpret effects of intercurrent events and missing data. Int J Obes (Lond). 2021 May;45(5):923-933. doi: 10.1038/s41366-020-00733-x. Epub 2021 Jan 18. PMID 33462358
- [Background] Yang X, Gong Y, Waheed N, March K, Bian J, Hogan WR, Wu Y. Identifying Cancer Patients at Risk for Heart Failure Using Machine Learning Methods. AMIA Annu Symp Proc. 2020 Mar 4;2019:933-941. eCollection 2019. PMID 32308890
- [Background] Zhang D, Advani S, Huchko M, Braithwaite D. Impact of healthcare access and HIV testing on utilisation of cervical cancer screening among US women at high risk of HIV infection: cross-sectional analysis of 2016 BRFSS data. BMJ Open. 2020 Jan 6;10(1):e031823. doi: 10.1136/bmjopen-2019-031823. PMID 31911515
- [Background] Pearl RL, Wadden TA, Tronieri JS, Berkowitz RI, Chao AM, Alamuddin N, Leonard SM, Carvajal R, Bakizada ZM, Pinkasavage E, Gruber KA, Walsh OA, Alfaris N. Short- and Long-Term Changes in Health-Related Quality of Life with Weight Loss: Results from a Randomized Controlled Trial. Obesity (Silver Spring). 2018 Jun;26(6):985-991. doi: 10.1002/oby.22187. Epub 2018 Apr 20. PMID 29676530
- [Background] Cessna JM, Jim HS, Sutton SK, Asvat Y, Small BJ, Salsman JM, Zachariah B, Fishman M, Field T, Fernandez H, Perez L, Jacobsen PB. Evaluation of the psychometric properties of the PROMIS Cancer Fatigue Short Form with cancer patients. J Psychosom Res. 2016 Feb;81:9-13. doi: 10.1016/j.jpsychores.2015.12.002. Epub 2015 Dec 11. PMID 26800633
- [Background] Cella D, Lai JS, Jensen SE, Christodoulou C, Junghaenel DU, Reeve BB, Stone AA. PROMIS Fatigue Item Bank had Clinical Validity across Diverse Chronic Conditions. J Clin Epidemiol. 2016 May;73:128-34. doi: 10.1016/j.jclinepi.2015.08.037. Epub 2016 Mar 3. PMID 26939927
- [Background] Cook KF, Bamer AM, Roddey TS, Kraft GH, Kim J, Amtmann D. A PROMIS fatigue short form for use by individuals who have multiple sclerosis. Qual Life Res. 2012 Aug;21(6):1021-30. doi: 10.1007/s11136-011-0011-8. Epub 2011 Sep 17. PMID 21927914
- [Background] Vitolins MZ, Blackwell CS, Katula JA, Isom SP, Case LD. Long-term Weight Loss Maintenance in the Continuation of a Randomized Diabetes Prevention Translational Study: The Healthy Living Partnerships to Prevent Diabetes (HELP PD) Continuation Trial. Diabetes Care. 2019 Sep;42(9):1653-1660. doi: 10.2337/dc19-0295. Epub 2019 Jul 11. PMID 31296648
- [Background] Schalet BD, Pilkonis PA, Yu L, Dodds N, Johnston KL, Yount S, Riley W, Cella D. Clinical validity of PROMIS Depression, Anxiety, and Anger across diverse clinical samples. J Clin Epidemiol. 2016 May;73:119-27. doi: 10.1016/j.jclinepi.2015.08.036. Epub 2016 Feb 27. PMID 26931289
- [Background] Hanish AE, Lin-Dyken DC, Han JC. PROMIS Sleep Disturbance and Sleep-Related Impairment in Adolescents: Examining Psychometrics Using Self-Report and Actigraphy. Nurs Res. 2017 May/Jun;66(3):246-251. doi: 10.1097/NNR.0000000000000217. PMID 28448375
- [Background] Kuo HK, Leveille SG, Yu YH, Milberg WP. Cognitive function, habitual gait speed, and late-life disability in the National Health and Nutrition Examination Survey (NHANES) 1999-2002. Gerontology. 2007;53(2):102-10. doi: 10.1159/000096792. Epub 2006 Nov 6. PMID 17090975
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Rantanen T, Guralnik JM, Foley D, Masaki K, Leveille S, Curb JD, White L. Midlife hand grip strength as a predictor of old age disability. JAMA. 1999 Feb 10;281(6):558-60. doi: 10.1001/jama.281.6.558. PMID 10022113
- [Background] Mendoza TR, Williams LA, Shi Q, Wang XS, Bamidele O, Woodruff JF, Cleeland CS. The Treatment-induced Neuropathy Assessment Scale (TNAS): a psychometric update following qualitative enrichment. J Patient Rep Outcomes. 2020 Feb 19;4(1):15. doi: 10.1186/s41687-020-0180-8. PMID 32076879
- [Background] Voorrips LE, Ravelli AC, Dongelmans PC, Deurenberg P, Van Staveren WA. A physical activity questionnaire for the elderly. Med Sci Sports Exerc. 1991 Aug;23(8):974-9. PMID 1956274
- [Background] Brady MJ, Cella DF, Mo F, Bonomi AE, Tulsky DS, Lloyd SR, Deasy S, Cobleigh M, Shiomoto G. Reliability and validity of the Functional Assessment of Cancer Therapy-Breast quality-of-life instrument. J Clin Oncol. 1997 Mar;15(3):974-86. doi: 10.1200/JCO.1997.15.3.974. PMID 9060536
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Block G, Gillespie C, Rosenbaum EH, Jenson C. A rapid food screener to assess fat and fruit and vegetable intake. Am J Prev Med. 2000 May;18(4):284-8. doi: 10.1016/s0749-3797(00)00119-7. PMID 10788730
- [Background] Sociali G, Grozio A, Caffa I, Schuster S, Becherini P, Damonte P, Sturla L, Fresia C, Passalacqua M, Mazzola F, Raffaelli N, Garten A, Kiess W, Cea M, Nencioni A, Bruzzone S. SIRT6 deacetylase activity regulates NAMPT activity and NAD(P)(H) pools in cancer cells. FASEB J. 2019 Mar;33(3):3704-3717. doi: 10.1096/fj.201800321R. Epub 2018 Dec 4. PMID 30514106
- [Background] Park HS, Park JY, Yu R. Relationship of obesity and visceral adiposity with serum concentrations of CRP, TNF-alpha and IL-6. Diabetes Res Clin Pract. 2005 Jul;69(1):29-35. doi: 10.1016/j.diabres.2004.11.007. Epub 2004 Dec 30. PMID 15955385
- [Background] Lerner L, Hayes TG, Tao N, Krieger B, Feng B, Wu Z, Nicoletti R, Chiu MI, Gyuris J, Garcia JM. Plasma growth differentiation factor 15 is associated with weight loss and mortality in cancer patients. J Cachexia Sarcopenia Muscle. 2015 Dec;6(4):317-24. doi: 10.1002/jcsm.12033. Epub 2015 Apr 30. PMID 26672741
- [Background] Ortega MS, Wohlgemuth S, Tribulo P, Siqueira LG, Cole JB, Hansen PJ. A single nucleotide polymorphism in COQ9 affects mitochondrial and ovarian function and fertility in Holstein cows. Biol Reprod. 2017 Mar 1;96(3):652-663. doi: 10.1093/biolre/iox004. PMID 28339599
- [Background] Suresh K. An overview of randomization techniques: An unbiased assessment of outcome in clinical research. J Hum Reprod Sci. 2011 Jan;4(1):8-11. doi: 10.4103/0974-1208.82352. PMID 21772732
- [Background] Moerbeek M. Optimal allocations for two treatment comparisons within the proportional odds cumulative logits model. PLoS One. 2021 Apr 21;16(4):e0250119. doi: 10.1371/journal.pone.0250119. eCollection 2021. PMID 33882086
- [Background] Fielding RA, Rejeski WJ, Blair S, Church T, Espeland MA, Gill TM, Guralnik JM, Hsu FC, Katula J, King AC, Kritchevsky SB, McDermott MM, Miller ME, Nayfield S, Newman AB, Williamson JD, Bonds D, Romashkan S, Hadley E, Pahor M; LIFE Research Group. The Lifestyle Interventions and Independence for Elders Study: design and methods. J Gerontol A Biol Sci Med Sci. 2011 Nov;66(11):1226-37. doi: 10.1093/gerona/glr123. Epub 2011 Aug 8. PMID 21825283
- [Background] LIFE Study Investigators; Pahor M, Blair SN, Espeland M, Fielding R, Gill TM, Guralnik JM, Hadley EC, King AC, Kritchevsky SB, Maraldi C, Miller ME, Newman AB, Rejeski WJ, Romashkan S, Studenski S. Effects of a physical activity intervention on measures of physical performance: Results of the lifestyle interventions and independence for Elders Pilot (LIFE-P) study. J Gerontol A Biol Sci Med Sci. 2006 Nov;61(11):1157-65. doi: 10.1093/gerona/61.11.1157. PMID 17167156
- [Background] American College of Sports Medicine; Chodzko-Zajko WJ, Proctor DN, Fiatarone Singh MA, Minson CT, Nigg CR, Salem GJ, Skinner JS. American College of Sports Medicine position stand. Exercise and physical activity for older adults. Med Sci Sports Exerc. 2009 Jul;41(7):1510-30. doi: 10.1249/MSS.0b013e3181a0c95c. PMID 19516148
- [Background] Nelson ME, Rejeski WJ, Blair SN, Duncan PW, Judge JO, King AC, Macera CA, Castaneda-Sceppa C. Physical activity and public health in older adults: recommendation from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1435-45. doi: 10.1249/mss.0b013e3180616aa2. PMID 17762378
- [Background] Conroy MB, McTigue KM, Bryce CL, Tudorascu D, Gibbs BB, Arnold J, Comer D, Hess R, Huber K, Simkin-Silverman LR, Fischer GS. Effect of Electronic Health Record-Based Coaching on Weight Maintenance: A Randomized Trial. Ann Intern Med. 2019 Dec 3;171(11):777-784. doi: 10.7326/M18-3337. Epub 2019 Nov 12. PMID 31711168
- [Background] Baecke JA, Burema J, Frijters JE. A short questionnaire for the measurement of habitual physical activity in epidemiological studies. Am J Clin Nutr. 1982 Nov;36(5):936-42. doi: 10.1093/ajcn/36.5.936. PMID 7137077
- [Background] Breteler MJ, Janssen JH, Spiering W, Kalkman CJ, van Solinge WW, Dohmen DA. Measuring Free-Living Physical Activity With Three Commercially Available Activity Monitors for Telemonitoring Purposes: Validation Study. JMIR Form Res. 2019 Apr 24;3(2):e11489. doi: 10.2196/11489. PMID 31017587
- [Background] Fuller D, Colwell E, Low J, Orychock K, Tobin MA, Simango B, Buote R, Van Heerden D, Luan H, Cullen K, Slade L, Taylor NGA. Reliability and Validity of Commercially Available Wearable Devices for Measuring Steps, Energy Expenditure, and Heart Rate: Systematic Review. JMIR Mhealth Uhealth. 2020 Sep 8;8(9):e18694. doi: 10.2196/18694. PMID 32897239
- [Background] Yang Y, Gharaibeh RZ, Newsome RC, Jobin C. Amending microbiota by targeting intestinal inflammation with TNF blockade attenuates development of colorectal cancer. Nat Cancer. 2020 Jul;1(7):723-734. doi: 10.1038/s43018-020-0078-7. Epub 2020 Jun 22. PMID 33768208
- [Background] Perri MG, Anton SD, Durning PE, Ketterson TU, Sydeman SJ, Berlant NE, Kanasky WF Jr, Newton RL Jr, Limacher MC, Martin AD. Adherence to exercise prescriptions: effects of prescribing moderate versus higher levels of intensity and frequency. Health Psychol. 2002 Sep;21(5):452-8. PMID 12211512
- [Background] Duncan GE, Anton SD, Sydeman SJ, Newton RL Jr, Corsica JA, Durning PE, Ketterson TU, Martin AD, Limacher MC, Perri MG. Prescribing exercise at varied levels of intensity and frequency: a randomized trial. Arch Intern Med. 2005 Nov 14;165(20):2362-9. doi: 10.1001/archinte.165.20.2362. PMID 16287765